CLINICAL TRIAL: NCT02716025
Title: Serum Zinc, Peptic Ulcer Disease and H. Pylori Infection
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Abdelhakam, Assistant Professor, Ain Shams University
Other Study IDs: 811
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Peptic Ulcer Disease
MeSH Terms: conditions — Peptic Ulcer | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Case Group
  Interventions: Procedure: Upper gastrointestinal endoscopy
- Control Group

INTERVENTIONS:
Procedure: Upper gastrointestinal endoscopy — Thorough examination of the esophagus, stomach and duodenum to the second part was done to all patients using Olympus CV-150 or Pentax EPM-3500.
  Groups: Case Group

SUMMARY:
Fifty consecutive patients with symptoms suggestive of peptic ulcer disease were included. All underwent complete clinical evaluation, laboratory investigations, upper gastrointestinal endoscopy and rapid urease test. Measurement of serum zinc level was done for all the included patients in addition to twenty five age and sex matched healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms suggestive of peptic ulcer disease like epigastric pain, dyspepsia, heartburn

Exclusion Criteria:

* Patients who received zinc supplementation, proton pump inhibitors (PPI), non-steroidal anti-inflammatory drugs (NSAIDs)
* Those presented with hematemesis or melena
* Those with chronic liver disease, renal failure, malabsorption or previous gastric surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with symptoms suggestive of peptic ulcer disease like epigastric pain, dyspepsia, heartburn who were candidates for upper gastrointestinal endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Detection of positive upper GIT endoscopic findings | upon endoscopy